CLINICAL TRIAL: NCT06440850
Title: A Pilot Clinical Trial of Vemurafenib and Cobimetinib as a Redifferentiation Strategy in High-Risk, Radioactive Iodine (RAI) Naïve, BRAFV600E Mutated Differentiated Thyroid Carcinoma Patients Undergoing Initial RAI Therapy
Brief Title: Vemurafenib and Cobimetinib for the Treatment of Patients With High Risk Differentiated Thyroid Carcinoma With BRAFV600E Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21522; NCI-2024-02359 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21522 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-04-19; First posted 2024-06-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Gland Follicular Carcinoma; Thyroid Gland Oncocytic Carcinoma; Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Specimen Handling; cobimetinib; X-Rays; Iodine-131; Magnetic Resonance Spectroscopy; Thyrotropin Alfa; Glycoprotein Hormones, alpha Subunit; High-Energy Shock Waves; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vemurafenib and cobimetinib) (Experimental): Patients receive vemurafenib PO BID for 6 weeks and cobimetinib PO QD for 3 weeks, followed by 1 week off, and then continuing for 2 weeks. Patients then receive iodine 131 PO followed by 3 additional days of vemurafenib PO BID and cobimetinib PO QD. Patients receive thyrogen IM daily for 2 days followed by I-123 diagnostic scan during screening and on study. Patients also undergo MRI during screening, PET scan or CT scan and blood sample collection throughout the study and ultrasound imaging and I-131 whole body scan during follow up.
  Interventions: Procedure: Biospecimen Collection; Drug: Cobimetinib; Procedure: Computed Tomography; Procedure: Diagnostic Imaging; Procedure: I-131 Uptake Test; Radiation: Iodine I-131; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Recombinant Thyrotropin Alfa; Procedure: Ultrasound Imaging; Drug: Vemurafenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Diagnostic Imaging — Undergo I-123 diagnostic scan
  Other Names: Medical Imaging
Procedure: I-131 Uptake Test — Undergo I-131 whole body scan
  Other Names: I 131 Uptake; I-131 Uptake and Scan; Radioactive Iodine Uptake
Radiation: Iodine I-131 — Given PO
  Other Names: 131-Iodine; Bound Iodide I-131; I 131; I-131; Iodide I-131; Iodide, I-131; Iodine 131; Iodine-131; Iodotope; Iodotrope
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Recombinant Thyrotropin Alfa — Given IM
  Other Names: Recombinant Thyrotropin Alpha; Recombinant TSH Alpha; Thyrogen; Thyroid Stimulating Hormone Alpha; Thyrotropin Alfa; TSH-alpha
Procedure: Ultrasound Imaging — Undergo neck ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf

SUMMARY:
This phase II trial tests how well vemurafenib and cobimetinib work in treating patients with high risk differentiated thyroid carcinoma with BRAFV600E mutation, in preparation for radioactive iodine therapy. Vemurafenib and cobimetinib are used in patients whose cancer has a mutated (changed) form of a gene called BRAF. They are in a class of medications called kinase inhibitors. They work by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving vemurafenib and cobimetinib may work better to treat patients with high risk differentiated thyroid carcinoma with BRAFV600E mutation, in preparation for radioactive iodine therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The proportion of BRAF mutated high-risk differentiated thyroid carcinoma patients who achieve excellent or indeterminate response with vemurafenib and cobimetinib treatment prior to initial radioactive iodine (RAI) therapy as defined by American Thyroid Association guideline.

SECONDARY OBJECTIVES:

I. The proportion of patients who had significant change on their I-123 scan before and after the targeted therapy.

II. To evaluate the safety and tolerability as determined by adverse events related to vemurafenib and cobimetinib combination therapy.

III. To evaluate the efficacy of vemurafenib and cobimetinib in enhancing RAI avidity by assessing the progression-free survival.

IV. To evaluate the diagnostic and prognostic value of thyroglobulin level as determined by thyroglobulin changes associated with treatment response.

V. To evaluate the tumor molecular characteristics in treatment responders as compared to non-responders.

OUTLINE:

Patients receive vemurafenib orally (PO) twice per day (BID) for 6 weeks and cobimetinib PO once per day (QD) for 3 weeks, followed by 1 week off, and then continuing for 2 weeks. Patients then receive iodine 131 PO followed by 3 additional days of vemurafenib PO BID and cobimetinib PO QD. Patients receive thyrogen intramuscularly (IM) daily for 2 days followed by I-123 diagnostic scan during screening and on study. Patients also undergo magnetic resonance imaging (MRI) during screening, positron emission tomography (PET) scan or computed tomography (CT) scan and blood sample collection throughout the study and ultrasound imaging and I-131 whole body scan during follow up.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Willingness to be followed for about 14 months
* Males or females aged ≥ 18 years at the time of informed consent
* Patients with thyroid carcinoma of follicular origin (papillary, follicular or Hurthle cell)
* Known positive BRAFV600E mutation (determined on a previous analysis and/or on a representative formalin-fixed paraffin embedded (FFPE) tumor samples or on a biopsy sample)
* High risk for recurrence according to the American Thyroid Association (ATA) guideline defined as having one or more of the features below:

  * Gross extrathyroidal extension
  * FTC with extensive vascular invasion (> 4), although less likely to have BRAF mutation
  * PTC with vascular invasion
  * Advanced nodal disease of (any node >3 cm, > 4 nodes, or extra-nodal extension)
  * BRAF+TERT promoter mutation
  * Post op thyroglobulin (TG) suggestive of distant metastasis
  * Distant metastatic sites (only for exploratory arm)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Blood pressure (BP) ≤ 140/90 mm Hg at screening with or without antihypertensive medications and no change in antihypertensive medications within 1 week prior to treatment start
* Creatinine clearance ≥ 50 mL/min according to the Cockcroft and Gault formula
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100 x 109/L
* Normal blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤ 1.5
* Bilirubin ≤ 1.5 × upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome
* Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 × ULN (≤ 5 × ULN if subject has liver metastases)
* Women of childbearing potential must have a negative urine or serum β-HCG pregnancy test within 7 days prior to the administration of the first study treatment
* Agreement by women of childbearing potential (WOCBP) and males of childbearing potential* to use an effective** method of birth control** for at least 3 months prior to screening through 1 year of study follow-up.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

    * Effective birth control defined as hormonal and/or barrier contraception
* Non-English speaking persons and adults lacking capacity to consent are not excluded from participation

Exclusion Criteria:

* Prior RAI treatment
* Prior anti-BRAF, anti-MEK treatment such as sorafenib, dabrafenib, vemurafenib, encorafenib, binimetinib, cobimetinib, trametinib, d selumitinib and other TKIs like, lenvatinib, sunitinib, axitinib, cabozantenib, vandatinib, pazopanib use
* Low to intermediate risk differentiated thyroid cancer (DTC) cases (not having the high-risk features as described above)
* RAI contraindication
* Undifferentiated or Medullary (MTC) carcinoma of the thyroid
* Major surgery within 4 weeks prior to the first dose of treatment
* Subjects having > 1 + proteinuria on urine dipstick testing will undergo 24 h urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥ 1 g/24 h will be ineligible
* Need for locoregional treatment such as surgery, external beam radiation or thermoablation at inclusion
* External beam radiation, for thyroid cancer, <4 weeks prior initiation of treatment
* Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of the drugs
* History of congestive heart failure greater or equal to than New York Heart association (NYHA) Class II, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of treatment, or cardiac arrhythmia associated with significant cardiovascular impairment and uncontrolled hypertension
* Electrocardiogram (ECG) with QT interval (QTc) interval ≥ 480 msec
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 2 months prior to the first dose of treatment and any other active bleeding, coagulopathy or pathologic condition that would confer a high risk of bleeding
* Active infection requiring systemic therapy
* Active malignancy (except for DTC, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or bladder) within the past 24 months
* Any history of or concomitant medical condition that, in the opinion of the investigator, would compromise subject's ability to safely complete the protocol
* Females who are pregnant or breastfeeding
* Patients with an injection of radio-contrast agent within 12 weeks prior to enrollment (can be enrolled after 12 weeks)
* Previous history of retinal vein occlusion
* Previous history of central serious retinopathy
* Known hypersensitivity to the study drugs or to any of the excipients
* Any other condition (including psychosocial condition) that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Any other condition that would confound study results
* Noncompliance
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Patients who achieve excellent or indeterminate response with vemurafenib and cobimetinib treatment prior to radioactive iodine therapy | Up to completion of 6 week vemurafenib and cobimetinib therapy
  Excellent and indeterminate responses are defined by 2015 American Thyroid Association Management Guildelines for Differentiated Thyroid Cancer:
  * Excellent: Negative imaging and either suppresed thyroglobulin < 0.2 ng/mL or TSH-stimulated thyroglobulin < 1 ng/mL
  * Indeterminate: Nonspecific findings on imaging studies, faint uptake in thyroid bed on RAI scans, nonstimulated thyroglobulin detectable, but <1 ng/mL, stimulated thyroglobulin detectable but <10 ng/mL or thyroglobulin antibodies stable or declining in the absence of structural or functional disease

SECONDARY OUTCOMES:
Proportion of patients who achieve increased iodine incorporation to a predicted lesion absorbed dose of 2000 cGy with I-131 dose of ≤ 300 mCi | Up to completion of 6 week vemurafenib and cobimetinib therapy
Incidence of treatment related adverse events | Up to completion of 6 week vemurafenib and cobimetinib therapy and 3 days of post-radioactive iodine therapy
  Will be summarized by type, severity (by Common Terminology Criteria for Adverse Events version 5.0 and nadir or maximum values for lab measures), date of onset, duration, reversibility, and attribution.
Progression free survival | Up to one year after treatment
  From initiation of study therapy to the first observation of disease relapse/progression or death from any cause, whichever occurs first.
Changes in thyroglobulin levels | Baseline, 3, 6, 9, months post-treatment up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Sasan Fazeli, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States